CLINICAL TRIAL: NCT02444754
Title: Patient Experience Protocol (PEP): A Pilot Study of Underserved Populations at the Comprehensive Cancer Center of Wake Forest University (CCCWFU)
Brief Title: Attitudes and Knowledge Regarding Clinical Trials in Underserved Populations Receiving Care at the Comprehensive Cancer Center of Wake Forest University
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00032590; NCI-2015-00685 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01215 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health services research (surveys, questionnaires): Patients complete survey items across a number of domains (patient characteristics, access to health care, perceived quality of care, clinical trial knowledge and attitudes, and cancer related health needs). Patients also complete questionnaires to obtain demographics information including age, education, race and ethnicity, marital status, employment status, insurance coverage, and income, as well as health status/indicators. Cancer-related characteristics, including diagnosis, stage, time since diagnosis, and treatments received are obtained self-report and patients' medical records.
  Interventions: Other: Medical Chart Review; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Medical Chart Review — Obtain medical data
  Other Names: Chart Review
Other: Questionnaire Administration — Complete demographics questionnaires
Other: Survey Administration — Complete surveys

SUMMARY:
This pilot research trial studies minority patients receiving care at the Comprehensive Cancer Center of Wake Forest University (CCCWFU) to see what their attitudes are regarding the healthcare they receive and how much they know about clinical trials. Clinical trials are an important way to test healthcare treatments and need diverse participants to be most effective. Studying what minority patients think about healthcare and clinical trials may help researchers learn more about why minorities are less likely to enroll in clinical trials and create programs to help increase their enrollment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe perceived quality of care received in the CCCWFU adult oncology clinics by patients belonging to one of the racial/ethnic minority and underserved populations (Hispanic/Latino, Black/African American, rural, uninsured, or young adult).

II. To describe cancer-related health needs of racial/ethnic minority and underserved patients in the CCCWFU adult oncology clinics.

III. To describe attitudes towards, and knowledge regarding, clinical trials in racial/ethnic minority and underserved patients treated in the CCCWFU adult oncology clinics.

SECONDARY OBJECTIVES:

I. To compare levels of perceived quality of care, cancer-related health needs and attitudes towards and knowledge of clinical trials in racial/ethnic minority and underserved patients to a comparison group of non-minority/underserved patients treated in the CCCWFU adult oncology clinics.

II. To describe perceived quality of care received in the CCCWFU adult oncology clinics, cancer-related health needs, and attitudes towards, and knowledge regarding clinical trials by elderly patients.

OUTLINE:

Patients complete survey items across a number of domains (patient characteristics, access to health care, perceived quality of care, clinical trial knowledge and attitudes, and cancer related health needs). Patients also complete questionnaires to obtain demographics information including age, education, race and ethnicity, marital status, employment status, insurance coverage, and income, as well as health status/indicators. Cancer-related characteristics, including diagnosis, stage, time since diagnosis, and treatments received are obtained self-report and patients' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a diagnosis of a malignant cancer
* Patients belonging to one of the minority/underserved populations: self-reported Hispanic/Latino or Black/African American, rural, uninsured, or young adult (ages 18-39) at the time of diagnosis, or are a randomly sampled patient with an upcoming scheduled appointment at CCCWFU that does not meet the definition of underserved for this study
* Patients who have a scheduled outpatient appointment physically located at a CCCWFU adult oncology clinic (main medical campus) and have completed at least three outpatient medical appointments at CCCWFU in the adult oncology clinics

Exclusion Criteria:

* Patients who receive their cancer care in clinics outside of adult oncology at CCCWFU
* Patients receiving care at the CCCWFU adult oncology clinics for screening, diagnostic or non-cancer related reasons only
* Unable or unwilling to consent or complete the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have received a diagnosis of a malignant cancer belonging to one of the minority/underserved populations.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2016-01; Primary Completion 2019-09-25 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Attitudes towards and knowledge regarding clinical trials | Baseline
  Descriptive statistics will be used to summarize patient attitudes towards and knowledge of clinical trials for each underserved group and for the elderly using means and standard deviations for continuous variables and frequencies for categorical variables.
Cancer-related health needs | Baseline
  Descriptive statistics will be used to summarize cancer-related health needs for each underserved group means and standard deviations for continuous variables and frequencies for categorical variables.
Perceived quality of care | Baseline
  Descriptive statistics will be used to summarize perceived quality of care for each underserved group using means and standard deviations for continuous variables and frequencies for categorical variables.

SECONDARY OUTCOMES:
Attitudes towards and knowledge regarding clinical trials | Baseline
  An ANOVA model will be used for continuous outcomes and a logistic model will be used for dichotomous outcomes with group (each underserved population or the comparison group) as the primary predictor to evaluate if the outcomes differ by group, utilizing contrasts to compare the underserved groups to each other, and the underserved groups as a whole to the comparison group. An overall alpha level of 0.05 will be used to indicate statistical significance for the comparison of the underserved group to the comparison group.
Attitudes towards and knowledge regarding clinical trials by the elderly | Baseline
  Descriptive statistics will be used to summarize attitudes towards and knowledge regarding clinical trials for the elderly using means and standard deviations for continuous variables and frequencies for categorical variables.
Cancer-related health needs by elderly patients | Baseline
  Descriptive statistics will be used to summarize cancer-related health needs for the elderly using means and standard deviations for continuous variables and frequencies for categorical variables.
Cancer-related needs | Baseline
  An ANOVA model will be used for continuous outcomes and a logistic model will be used for dichotomous outcomes with group (each underserved population or the comparison group) as the primary predictor to evaluate if the outcomes differ by group, utilizing contrasts to compare the underserved groups to each other, and the underserved groups as a whole to the comparison group. An overall alpha level of 0.05 will be used to indicate statistical significance for the comparison of the underserved group to the comparison group.
Perceived quality of care | Baseline
  An analysis of variance (ANOVA) model will be used for continuous outcomes and a logistic model will be used for dichotomous outcomes with group (each underserved population or the comparison group) as the primary predictor to evaluate if the outcomes differ by group, utilizing contrasts to compare the underserved groups to each other, and the underserved groups as a whole to the comparison group. An overall alpha level of 0.05 will be used to indicate statistical significance for the comparison of the underserved group to the comparison group.
Perceived quality of care received by elderly patients | Baseline
  Descriptive statistics will be used to summarize perceived quality of care for the elderly using means and standard deviations for continuous variables and frequencies for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Ruiz, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States